CLINICAL TRIAL: NCT02740231
Title: A Two-stage 6-month Multicentre, Randomised, Double-blind, Controlled Study on the Safety and Efficacy Intra-articular Administration of JTA-004 in Patients With Symptomatic Knee Osteoarthritis
Brief Title: A Study on Visco-antalgic Intra-articular Administration in Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: JTA-KOA1
Record Dates: First submitted 2016-04-13; First posted 2016-04-15 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: Knee Osteoarthritis
Keywords: viscosupplement; osteoarthritis; knee; intra-articular injection; arthritis; degenerative
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reference product (Active Comparator): Hylan G-F 20
  Interventions: Device: Reference product intra-articular injection
- JTA-004 50 (2 ml) (Experimental): Sodium hyaluronate, plasma proteins and clonidine
  Interventions: Drug: JTA-004 intra-articular injection
- JTA-004 50 (4 ml) (Experimental): Sodium hyaluronate, plasma proteins and clonidine
  Interventions: Drug: JTA-004 intra-articular injection
- JTA-004 100 (2 ml) (Experimental): Sodium hyaluronate, plasma proteins and clonidine
  Interventions: Drug: JTA-004 intra-articular injection

INTERVENTIONS:
Drug: JTA-004 intra-articular injection — Each patient will undergo a single injection of JTA-004 into the knee joint
  Arms: JTA-004 100 (2 ml); JTA-004 50 (2 ml); JTA-004 50 (4 ml)
Device: Reference product intra-articular injection — Each patient will undergo a single injection of Reference product into the knee joint
  Arms: Reference product

SUMMARY:
Osteoarthritis (OA) is the most common joint disease affecting millions of people around the world, for which there is unfortunately no cure. Among existing therapies, viscosupplementation, i.e., the injection of hyaluronic acid into the joint, has an established place in the symptomatic treatment of knee OA.

The present Phase IIb/III aiming to assess the safety and efficacy of JTA-004 is organized in two phases. With results obtained in the first phase the best dose of JTA-004 is determined, and the efficacy of the selected dose will then be confirmed in the second phase.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Diagnosed with primary knee osteoarthritis, fulfilling the following American College of Rheumatology (ACR) criteria at the target knee:

  * Pain ≥ 40 mm on a 0-100 mm VAS during the 3 days preceding the date of the screening visit
  * Morning stiffness not exceeding 30 minutes
  * Kellgren-Lawrence grade II or III
* Insufficient / failed response to analgesic and / or NSAIDs
* No physical therapy of the knee, and knee braces for the entire duration of study
* Ability to provide a written, dated, and signed informed consent prior to any study related procedure, and to understand and comply with study requirements

Exclusion Criteria:

Current symptoms and/or signs related to the disease under study:

* Isolated symptomatic femoropatellar OA of the target knee
* History of trauma or surgery or arthroscopy at the target knee within 6 months before inclusion
* Concomitant inflammatory disease or other condition affecting the joints (e.g., rheumatoid arthritis, septic arthritis, inflammatory joint disease, metabolic bone disease, psoriasis, gout, microcrystalline arthropathies/chondrocalcinosis, Paget's disease)
* Any musculoskeletal condition (such as hip osteoarthritis, amputation, neurologic disorder) that would impede measurement of efficacy at target knee
* Target knee prosthesis planned within 12 months after the Screening Visit

Current or previous diagnoses, signs and/or symptoms:

* Uncontrolled diabetes mellitus, end-stage hepatic or renal disease
* Current (or within the last 5 years prior to entering the study) history of solid or haematological neoplasia or bone marrow transplantation (except for basal cell carcinoma and completely excised squamous cell carcinoma)
* Other severe acute or chronic medical or psychiatric conditions or pre-dispositions or laboratory abnormalities, as judged by the Investigator
* Current or past history of coagulation disorders, as judged by the Investigator
* Hypersensitivity to any components of HA-based injection products
* History of hypersensitivity to human biological material including blood and blood derived products, potential excipients and residues from manufacturing process documented clinically or by laboratory tests
* Hypersensitivity to avian proteins
* Life expectancy less than 6 months

Current or previous treatment:

* Participation in another clinical study within 6 months prior to Screening
* Patients previously treated with JTA-004
* Treatment:

  * Within 6 months prior to Screening: intra-articular hyaluronic acid injection at the target knee
  * Within 2 months prior to Screening: intra-articular glucocorticoids at the target knee
* Current chemo-, radio- or immuno-cancer-therapy or immunosuppressive therapy
* Current anti-hypertensive medication the effects of which are known to be potentiated by a single dose of clonidine
* Current (or within 6 months prior to Screening) illicit drug abuse

Safety aspects concerning female subjects of childbearing potential:

* Females who are pregnant, lactating or woman with childbearing potential (last menstrual bleeding less than 12 months ago) unwilling to use medically acceptable contraception, or women with childbearing potential unwilling to perform a pregnancy test before administration of study treatment.

Other exclusion criteria:

* Body Mass Index (BMI) of 35 kg/m2 or greater

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

REFERENCES:
- [Derived] Bettonville M, Leon M, Margaux J, Urbin-Choffray D, Theunissen E, Besse-Hammer T, Fortems Y, Verlinden S, Godeaux O, Delmarcelle AS, Kaux JF. Safety and efficacy of a single intra-articular injection of a novel enhanced protein solution (JTA-004) compared to hylan G-F 20 in symptomatic knee osteoarthritis: a randomized, double-blind, controlled phase II/III study. BMC Musculoskelet Disord. 2021 Oct 19;22(1):888. doi: 10.1186/s12891-021-04750-3. PMID 34666767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From the patients enrolled in the study at Visit #1 (screening visit), 173 patients were randomized just before Visit #2 (within 6 weeks after confirmation of eligibility). During visit #2, a total of 164 patients were treated (41 subject in each treatment group) and included in the FAS.
  9 randomized patients were not treated.
Period: Overall Study
Arm/Group | Reference Product | JTA-004 50 (2 ml) | JTA-004 50 (4 ml) | JTA-004 100 (2 ml)
Started | 41 | 41 | 41 | 41
Completed | 39 | 35 | 40 | 33
Not Completed | 2 | 6 | 1 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 4
Not completed — Lost to Follow-up | 1 | 3 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference Product | JTA-004 50 (2 ml) | JTA-004 50 (4 ml) | JTA-004 100 (2 ml) | Total
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (7.7) | 64.2 (8.0) | 62.9 (7.2) | 61.7 (7.0) | 62.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 27 | 24 | 112
  Male | 11 | 10 | 14 | 17 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 41 | 41 | 41 | 41 | 164
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (4.2) | 29.0 (3.9) | 28.0 (3.6) | 29.6 (3.5) | 28.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in WOMAC VA3.1 Pain Subscale Score at Month 6
Description: The primary endpoint is the Western Ontario McMaster universities (WOMAC®) VA3.1 Pain Subscale (subscale A): the individual changes in WOMAC® VA3.1 Pain Subscale Score between Baseline and Month 6 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group.
  Results are expressed as "adjusted mean" based on the model used for group comparison.
  WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity ans osteonecrosis symptoms. The WOMAC® Index Pain Subscale (VAS format) was used. The VAS score was determined by measuring in millimetres from the left-hand end of the line to the point that the patient marks (0-100 mm) for 5 questions. Results are summed and normalized on a 100 mm scale: 0 represents no knee pain and 100 extreme knee pain.
Time Frame: Baseline and 6 months
Population: The primary efficacy parameter results were evaluated on JTA-004 100 (2 mL) (the most effective strength) and reference group only.
  From the 41 patients treated per group, pain subscale evaluation was not performed at 6 months for 6 patients from JTA-004 100 (2 mL) and 2 patients from Reference product group due to patient discontinuation.
  Statistical analysis was performed on the Full Analysis Set (FAS) (= all randomized and treated patients).
Measure: Mean (Standard Error); unit: mm
Arm/Group | JTA-004 100 (2 mL) | Reference Product
Number analyzed (Participants) | 35 | 39
mm | -23.6 (4.6) | -14.1 (4.3)
Statistical Analysis 1: Comparison: JTA-004 100 (2 mL) vs Reference Product; The primary endpoint is the WOMAC® VA3.1 Pain Subscale (subscale A): the individual changes in WOMAC® VA3.1 Pain Subscale Score between Baseline and Month 6 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group; Test type: Superiority; p = 0.141, ANCOVA — The threshold for statistical significance was p=0.05; Adjusted mean difference = -9.49, 95% CI 2-sided [-22.21 to 3.23], Standard Deviation 6.38 — Difference between groups JTA-004 100 (2mL) minus Reference - adjusted mean change

2. Secondary Outcome: WOMAC® Pain Subscale at Month 3
Description: The primary endpoint is the Western Ontario McMaster universities (WOMAC®) VA3.1 Pain Subscale (subscale A): the individual changes in WOMAC® VA3.1 Pain Subscale Score between Baseline and Month 3 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group.
  Results are expressed as "adjusted mean" based on the model used for group comparison.
  WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity ans osteonecrosis symptoms. The WOMAC® Index Pain Subscale (VAS format) was used. The VAS score was determined by measuring in millimetres from the left-hand end of the line to the point that the patient marks (0-100 mm) for 5 questions. Results are summed and normalized on a 100 mm scale: 0 represents no knee pain and 100 extreme knee pain.
Time Frame: Baseline and 3 months
Population: The secondary efficacy parameter results were evaluated on JTA-004 100 (2 mL) (the most effective strength) and reference group only.
  From the 41 patients treated per group, pain subscale evaluation at 3 month was not performed for 6 patients from JTA-004 100 (2 mL) and 1 patients from Reference product group due to patient discontinuation.
  Statistical analysis was performed on the Full Analysis Set (FAS) (= all randomized and treated patients).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 100 (2 mL) | Reference Product
Number analyzed (Participants) | 35 | 40
mm | -26.8 (3.9) | -15.1 (3.7)
Statistical Analysis 1: Comparison: JTA-004 100 (2 mL) vs Reference Product; Test type: Superiority; p = 0.038, ANCOVA — The threshold for statistical significance was p=0.05; Adjusted mean difference = -11.63, 95% CI 2-sided [-22.60 to -0.66], Standard Deviation 5.50 — Difference between groups JTA-004 100 (2mL) minus Reference

3. Secondary Outcome: WOMAC® Total Score Over Time
Description: The Western Ontario McMaster universities (WOMAC®) VA3.1 Total Score was used: the individual changes in WOMAC VA3.1 Total Score between Baseline and 2 weeks were calculated and compared by Mixed-Effect Model for Repeated Measurements, adjusted for baseline value, to the Reference group.
  Results are expressed as "adjusted mean" based on the model used for group comparison.
  WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity and osteonecrosis symptoms. The Total score (VAS format) was determined by measuring in millimetres from the left hand end of the line to the point that the patient marks (0-100 mm) for the pain (5 questions), stiffness (2 questions), and physical function (17 questions). Results are normalized on a 0-100 mm scale format. A higher score represents a higher degree of k
Time Frame: Baseline and 2 weeks
Population: The primary efficacy parameter results were evaluated on JTA-004 100 (2 mL) (the most effective strength) and reference group only.
  Full Analysis Set (FAS) = all randomized and treated patients
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 100 (2 mL) | Reference Product
Number analyzed (Participants) | 41 | 41
mm | -21.0 (3.1) | -19.5 (3.1)
Statistical Analysis 1: Comparison: JTA-004 100 (2 mL) vs Reference Product; Test type: Superiority; p = 0.997, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Adjusted mean difference = -1.48, 95% CI 2-sided [-12.70 to 9.74], Standard Deviation 4.35

4. Secondary Outcome: WOMAC® Total Score Over Time
Description: The Western Ontario McMaster universities (WOMAC®) VA3.1 Total Score was used: the individual changes in WOMAC VA3.1 Total Score between Baseline and Month 3 were calculated and compared by Mixed-Effect Model for Repeated Measurements, adjusted for baseline value, to the Reference group.
  Results are expressed as "adjusted mean" based on the model used for group comparison.
  WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity ans osteonecrosis symptoms. The Total score (VAS format) was determined by measuring in millimetres from the left hand end of the line to the point that the patient marks (0-100 mm) for the pain (5 questions), stiffness (2 questions), and physical function (17 questions). Results are normalized on a 0-100 mm scale format. A higher score represents a higher degree of knee disease severity.
Time Frame: Baseline and 3 months
Population: The primary efficacy parameter results were evaluated on JTA-004 100 (2 mL) (the most effective strength) and reference group only. From the 41 patients treated per group, total score evaluation was not performed at month 3 for 7 patients from JTA-004 100 (2 mL) group and 1 patient from Reference group due to discontinuation of patients and deviation (at least one subscale of Total score not evaluated) Full Analysis Set (FAS) (= all randomized and treated patients)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 100 (2 ml) | Reference Product
Number analyzed (Participants) | 34 | 40
mm | -22.3 (3.8) | -19.4 (3.6)
Statistical Analysis 1: Comparison: JTA-004 100 (2 ml) vs Reference Product; Test type: Superiority; p = 0.972, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Adjusted mean difference = -2.94, 95% CI 2-sided [-16.52 to 10.65], Standard Deviation 5.3

5. Secondary Outcome: WOMAC® Total Score Over Time
Description: The Western Ontario McMaster universities (WOMAC®) VA3.1 Total Score was used: the individual changes in WOMAC VA3.1 Total Score between Baseline and Month 6 were calculated and compared by Mixed-Effect Model for Repeated Measurements, adjusted for baseline value, to the Reference group.
  Results are expressed as "adjusted mean" based on the model used for group comparison.
  WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity ans osteonecrosis symptoms.The Total score (VAS format) was determined by measuring in millimetres from the left hand end of the line to the point that the patient marks (0-100 mm) for the pain (5 questions), stiffness (2 questions), and physical function (17 questions). Results are normalized on a 0-100 mm scale format. A higher score represents a higher degree of knee disease severity.
Time Frame: Baseline and 6 months
Population: The primary efficacy parameter results were evaluated on JTA-004 100 (2 mL) (the most effective strength) and reference group only. From the 41 patients treated per group, total score evaluation was not performed at month 6 for 6 patients from JTA-004 100 (2 mL) group and 2 patient from Reference group due to discontinuation of patients or deviation (at least one subscale of Total score not evaluated) Full Analysis Set (FAS) (= all randomized and treated patients)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 100 (2 ml) | Reference Product
Number analyzed (Participants) | 35 | 39
mm | -23.7 (4.3) | -16.5 (4.1)
Statistical Analysis 1: Comparison: JTA-004 100 (2 ml) vs Reference Product; Test type: Superiority; p = 0.599, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Adjusted mean difference = -7.17, 95% CI 2-sided [-22.28 to 7.94], Standard Deviation 5.96

6. Post Hoc Outcome: WOMAC® Total Score Over Time From Pooled JTA-004 Treatment Groups
Description: The Western Ontario McMaster universities (WOMAC®) VA3.1 Total Score was used: the individual changes in WOMAC VA3.1 Total Score between Baseline and Month 3 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group. Results are expressed as "adjusted mean" based on the model used for group comparison. WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity and osteonecrosis symptoms. The Total score (VAS format) was determined by measuring in mm from the left hand end of the line to the point that the patient marks (0-100 mm) for the pain (5 questions), stiffness (2 questions), and physical function (17 questions). Results are normalized on a 0-100 mm scale format. A higher score represents a higher degree of knee disease severity.
Time Frame: Baseline and 3 months
Population: A post-hoc analysis was conducted comparing pooled JTA-004 treated patients (all strengths) and patients treated with Reference product to complete the study and evaluate the efficacy of JTA-004 product versus Reference.
  At month 3, on the 41 patients treated per group, 3 patients from JTA 50 (2ml), 7 patients from JTA 100 (2 ml) and 1 patient from Reference were not analysed for total score due to patient discontinuation or deviation (at least one subscale not evaluated)
Measure: Mean (Standard Deviation); unit: mm
Groups:
- JTA-004 (All Strenghts): JTA-004 intra-articular injection: Each patient will undergo a single injection of JTA-004 into the knee joint
Arm/Group | JTA-004 (All Strenghts) | Reference Product
Number analyzed (Participants) | 113 | 40
mm | -26.3 (2.2) | -19.7 (3.7)
Statistical Analysis 1: Comparison: JTA-004 (All Strenghts) vs Reference Product; Test type: Superiority; p = 0.126, ANCOVA — The threshold for statistical significance was p=0.05; Adjusted mean difference = -6.62, Standard Deviation 4.3

7. Post Hoc Outcome: WOMAC® Total Score Over Time From Pooled JTA-004 Treatment Groups
Description: The Western Ontario McMaster universities (WOMAC®) VA3.1 Total Score was used: the individual changes in WOMAC Total Score between Baseline and Month 6 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group. Results are expressed as "adjusted mean" based on the model used for group comparison. WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity and osteonecrosis symptoms. The Total score (VAS format) was determined by measuring in millimetres from the left hand end of the line to the point that the patient marks (0-100 mm) for the pain (5 questions), stiffness (2 questions), and physical function (17 questions). Results are normalized on a 0-100 mm scale format. A higher score represents a higher degree of knee disease severity.
Time Frame: Baseline and 6 months
Population: A comparison of pooled JTA-004 treated patients (all strengths) vs Reference group was conducted to evaluate the efficacy of JTA-004 product versus Reference. At month 6, on the 41 patients treated per group, 5 patients JTA 50(2ml), 1 patient JTA 50 (4ml), 6 patients JTA 100 (2 ml) and 2 patients from Reference were not analysed for total score due to patient discontinuation or deviation (at least one subscale not evaluated) Full Analysis Set (FAS) (= all randomized and treated patients)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 (All Strenghts) | Reference Product
Number analyzed (Participants) | 111 | 39
mm | -26.2 (2.4) | -17.3 (4.1)
Statistical Analysis 1: Comparison: JTA-004 (All Strenghts) vs Reference Product; Test type: Superiority; p = 0.064, ANCOVA — The threshold for statistical significance was p=0.05; Adjusted mean difference = -8.88, Standard Deviation 4.76

8. Post Hoc Outcome: WOMAC® Pain Subscale Over Time From Pooled JTA-004 Treatment Groups
Description: The primary endpoint is the Western Ontario McMaster universities (WOMAC®) VA3.1 Pain Subscale A: the individual changes in WOMAC® Pain Subscale Score between Baseline and Month 3 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group. Results are expressed as "adjusted mean" based on the model used for group comparison. WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity ans osteonecrosis symptoms. The WOMAC® Index Pain Subscale (VAS format) was used. The VAS score was determined by measuring in millimetres from the left-hand end of the line to the point that the patient marks (0-100 mm) for 5 questions. Results are summed and normalized on a 100 mm scale: 0 represents no knee pain and 100 extreme knee pain.
Time Frame: Baseline and 3 months
Population: A comparison od pooled JTA-004 treated patients (all strengths) and Reference group was conducted to complete the study and evaluate the efficacy of JTA-004 product versus Reference. On the 41 patients treated per group, 2 patients from JTA 50 (2ml), 6 patients from JTA 100 (2 ml) and 1 patient from Reference were not analysed for total score due to patient discontinuation.
  Full Analysis Set (FAS) (= all randomized and treated patients)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 (All Strenghts) | Reference Product
Number analyzed (Participants) | 115 | 40
mm | -27.2 (2.2) | -16.4 (3.7)
Statistical Analysis 1: Comparison: JTA-004 (All Strenghts) vs Reference Product; Test type: Superiority; p = 0.014, ANCOVA; Adjusted mean difference = -10.79, Standard Deviation 4.35

9. Post Hoc Outcome: WOMAC® Pain Subscale Score Over Time From Pooled JTA-004 Treatment Groups
Description: The Western Ontario McMaster universities (WOMAC®) VA3.1 Total Score was used: the individual changes in WOMAC Total Score between Baseline and M6 were calculated and compared by analysis of covariance (ANCOVA), adjusted for baseline value, to the Reference group. Results are expressed as "adjusted mean" based on the model used for group comparison. WOMAC Osteoarthritis Index is a tri-dimensional, self-administered, patient-centred health status questionnaire for knee disease severity and osteonecrosis symptoms. . The Total score (VAS format) was determined by measuring in millimetres from the left hand end of the line to the point that the patient marks (0-100 mm) for the pain (5 questions), stiffness (2 questions), and physical function (17 questions). Results are normalized on a 0-100 mm scale format. A higher score represents a higher degree of knee disease severity.
Time Frame: Baseline and 6 months
Population: A comparison of pooled JTA-004 treated patients (all strengths) and Reference was conducted to evaluate the efficacy of JTA-004 product versus Reference. On the 41 patients treated per group, 5 patients from JTA 50 (2ml), 1 patient from JTA 50 (4ml), 6 patients from JTA 100 (2 ml) and 2 patients from Reference were not analysed for total score due to patient discontinuation Full Analysis Set (FAS) (= all randomized and treated patients)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | JTA-004 (All Strenghts) | Reference Product
Number analyzed (Participants) | 111 | 39
mm | -26.1 (2.4) | -15.6 (4.1)
Statistical Analysis 1: Comparison: JTA-004 (All Strenghts) vs Reference Product; Test type: Superiority; p = 0.030, ANCOVA — The threshold for statistical significance was p=0.05; Adjusted mean difference = -10.57, Standard Deviation 4.81

ADVERSE EVENTS:
Time Frame: 6 months post injection
Description: No death was reported during the study
Arm/Group | Reference Product | JTA-004 50 (2 ml) | JTA-004 50 (4 ml) | JTA-004 100 (2 ml)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/41 | 4/41 | 1/41 | 2/41
Other Adverse Events (participants affected / at risk) | 11/41 | 3/41 | 12/41 | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Product (N=41) | JTA-004 50 (2 ml) (N=41) | JTA-004 50 (4 ml) (N=41) | JTA-004 100 (2 ml) (N=41)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Barett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diaorrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Product (N=41) | JTA-004 50 (2 ml) (N=41) | JTA-004 50 (4 ml) (N=41) | JTA-004 100 (2 ml) (N=41)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Application Site Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conditions aggravated (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Delayed Recovery from Anesthesia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood and Creatine Phosphokinase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Amylase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Triglycerides Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Injection (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis Chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT02740231/Prot_SAP_000.pdf